CLINICAL TRIAL: NCT02309684
Title: The Clinical & Economic Evaluation of Bio-ConneKt® Wound Dressing in Treating Chronic Foot Ulcers (Diabetic and/or Venous Ulcers).
Brief Title: Bio-ConneKt Wound Dressing for Treatment of Chronic Leg Wounds: A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MLM Biologics Inc., (Industry)
Responsible Party: Sponsor
Other Study IDs: MLM1301
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Skin Ulcer
Keywords: Diabetic Foot Ulcer (DFU); Venous Leg Ulcer (VLU)
MeSH Terms: conditions — Skin Ulcer; Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population: Study population are subjects at least 18 years old and of any ethnic background with a full thickness diabetic foot ulcer or venous leg ulcer, where the ulcer has been diagnosed/present for greater than 4 weeks duration.

SUMMARY:
The purpose of this study is to assess the performance of the bio-ConneKt™ wound dressing and compare its performance with the standard of care at NFRMC Wound Therapy Services, for the treatment of chronic foot/leg ulcers (DFU/VLU) in a prospective single center open one-arm clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. A full thickness diabetic foot ulcer with a viable wound bed free of necrotic material (grade 1 on Wagner scale) or a venous leg ulcer confirmed with duplex ultrasound
2. The ulcer has been diagnosed/present for greater than 4 weeks duration.
3. Three or fewer ulcers separated by > 3.0 cm distance
4. Post-debridement, the ulcer size must be > 5 sq cm
5. Ankle / brachial index is between 0.7 to 1.2 and or one of the following must be present:

   1. transcutaneous partial pressure oxygen (TcPO2) > 30 mmHg at the ankle
   2. toe pressure of >40mm Hg or a Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic)
6. At least 18 years old
7. Able and willing to read and sign a voluntary written informed consent
8. Able and willing to attend scheduled follow-up visits and study related exams

Exclusion Criteria:

1. Greater than 30% reduction in wound size (DFU) or 20% reduction in VLU during first week of observation by the investigator
2. Ulcer with exposed tendon or bone
3. Gross clinical infection at the study ulcer site including cellulitis and osteomyelitis
4. Ulcer of a non-diabetic/non-venous pathophysiology (e.g., rheumatoid, radiation-related, and vasculitis related ulcers)
5. Known severe anemia
6. Known serum albumin < 2.5
7. Renal failure requiring dialysis
8. Rheumatoid arthritis (and other collagen vascular disease), vasculitis, sickle cell disease, HIV
9. Severe liver disease as defined by the treating physician or patient's primary care physician
10. Malignancy at or near the ulcer site
11. Any condition judged by the investigator that would cause the study to be detrimental to the patient
12. Presence of a hematology, clinical, chemistry or other test obtained within 7 days of screening that is outside the normal range for the laboratory and is determined to be clinically significant by the investigator
13. Received another investigational device or drug within 30 days of Day 0.
14. Radiation therapy, chemotherapy or immunosuppressive therapy within 30 days of enrollment
15. Received another allograft, autograft or xenograft within 30 days of the Day 0/
16. Known allergy to equine derived tissue
17. Alcohol or drug abuse, defined as current medical treatment for substance abuse
18. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 patients with DFU (n=10) and VLU (n=10) will be considered in this study if they sign the informed consent, and meet all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound closure | Weekly assessment up to 12 weeks
  Time to complete wound closure and percent wounds healed at 12 weeks

SECONDARY OUTCOMES:
Rate of Wound Closure | 4, 6, 12 & 24 weeks
  Mean and median wound size changes at 4, 6, 12 & 24 weeks, along with ulcer recurrence and/or device related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Elmer Croushore, MD, Principal Investigator — NFRMC Wound Therapy Services